CLINICAL TRIAL: NCT02770976
Title: Respiratory Pattern During Neurally Adjusted Ventilator Assist (NAVA) in Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inha University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: NAVA-03-INV
Record Dates: First submitted 2016-05-10; First posted 2016-05-12 (Estimated); Last update posted 2018-01-26 (Actual); Status verified 2018-01

CONDITIONS: Respiratory Distress Syndrome In Premature Infants; Preterm Infants
MeSH Terms: conditions — Respiratory Distress Syndrome In Premature Infants

ARMS (1):
- NAVA (Experimental): Seven increasing and decreasing NAVA levels (0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 3.5, 3.0, 2.5, 2.0, 1.5, 1.0 and 0.5 cmH2O/uV) will applied to 20 preterm infants each for 10 minutes.
  Interventions: Device: Increasing and decreasing NAVA levels with 10-min intervals

INTERVENTIONS:
Device: Increasing and decreasing NAVA levels with 10-min intervals

SUMMARY:
This study is to investigate the effect of a wide range of assistance levels on respiratory pattern, breathing variability including tidal volume and peak inspiratory pressure during neurally adjusted ventilatory assist (NAVA) in preterm infants. The investigators also aim to explore whether the effects of NAVA on the electrical activity of diaphragm (Edi) signal amplitude, work of breathing and comfort of preterm infants.

ELIGIBILITY:
Inclusion Criteria:

* preterm infants born before 36 weeks of gestational age
* who received mechanical ventilatory care through the endotracheal tube at least 24 hours for respiratory distress
* no use of anesthetics or analgetics

Exclusion Criteria:

* with major congenital anomalies (facial, gastrointestinal tract, cardiac, etc)
* with phrenic nerve palsy or injuries

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2016-05; Primary Completion 2017-03-09 (Actual); Study Completion 2017-03-09 (Actual)

PRIMARY OUTCOMES:
maximum Edi | the middle 2 minutes duration out of the total interval of 10 minutes
  mean of recorded maximum electrical activities in the middle 2 min duration out of the total 10 min period

SECONDARY OUTCOMES:
comfort score | the 5-min point in the total 10-min period
  calculated score of premature infant pain profile (PIPP) from the recorded video, heart rates and oxygen saturation
peak inspiratory pressure | the middle 2 minutes duration out of the total interval of 10 minutes
  mean of recorded peak inspiratory pressures in the middle 2 min duration out of the total 10 min period
tidal volume | the middle 2 minutes duration out of the total interval of 10 minutes
  mean of recorded expiratory tidal volumes in the middle 2 min duration out of the total 10 min period
inspiratory time in excess | the middle 2 minutes duration out of the total interval of 10 minutes
  mean of calculated excessive inspiratory times from the calculation ((ventilator pressurization time-neural inspiratory time)/neural inspiratory time) from the middle 2 min duration out of the total 10 min period
electrical time product | the middle 2 minutes duration out of the total interval of 10 minutes
  mean of calculated electrical time product from the middle 2 min duration out of the total 10 min period

CONTACTS AND LOCATIONS:
Locations (1):
- Inha University Hospital, Incheon, South Korea

REFERENCES:
- [Derived] Nam SK, Lee J, Jun YH. Neural feedback is insufficient in preterm infants during neurally adjusted ventilatory assist. Pediatr Pulmonol. 2019 Aug;54(8):1277-1283. doi: 10.1002/ppul.24352. Epub 2019 May 11. PMID 31077579